CLINICAL TRIAL: NCT03077243
Title: LCCC 1612: P53 Mutational Status and Circulating Free HPV DNA for the Management of HPV-associated Oropharyngeal Squamous Cell Cancers
Brief Title: P53 Mutational Status and cf HPV DNA for the Management of HPV-associated OPSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1612
Record Dates: First submitted 2017-01-30; First posted 2017-03-10 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms
Keywords: Human Papillomavirus; Oropharynx; Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma; Radiation Therapy; Chemotherapy; p16
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiotherapy and/or chemotherapy. (Experimental): Subjects with Oropharyngeal Squamous Cell Carcinoma receiving radiotherapy and/or chemotherapy.
  Interventions: Radiation: Intensity Modulated Radiotherapy (IMRT); Drug: Cisplatin (or alternative); Procedure: Assessment for surgical evaluation

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy (IMRT) — 60- 70 Gy at 2 Gy/fx
Drug: Cisplatin (or alternative) — The acceptable weekly chemotherapy regimens are Cisplatin 30 to 40 mg/m2 (first choice), Cetuximab 250mg/m2 (second choice), Carboplatin AUC 1.5 and paclitaxel 45 mg/m2 (third choice), Carboplatin AUC 3 (fourth choice). Chemotherapy will be given intravenously weekly during IMRT, 6 -7 total doses.
Procedure: Assessment for surgical evaluation — Decision for surgical evaluation will be based on the results of the PET/CT and clinical exam 10-16 weeks after CRT. Patients with a positive PET/CT scan will undergo surgical evaluation at the discretion of the surgeon. Patients with a negative PET/CT scan will be observed.

SUMMARY:
The primary objective of this study is to evaluate whether genomic based risk-stratification can be used in deciding whether to de-intensify in patients with Human Papillomavirus (HPV)-associated Oropharyngeal Squamous Cell Carcinoma (OPSCC) with > 10 pack years smoking history. Hypothesis: Patients with HPV-associated OPSCC, > 10 pack years smoking history, and non-mutated p53 will have similar 2 year progression-free survival (PFS) as patients with < 10 pack years smoking history.

DETAILED DESCRIPTION:
The proposed study is a follow-up study to LCCC 1120 and 1413. The investigators have shown that de-intensification is efficacious in these two phase II studies. A major question is whether the investigators can de-intensify in patients with HPV-associated oropharyngeal cancer who have smoking histories. The investigators' hypothesis is that genomic profiling of patients' tumors (specifically for p53 mutations) will help in triaging patients to de-intensification versus standard of care. Patients with HPV-associated OPSCC will be enrolled regardless of smoking history and p53 mutational status will be assessed in patients with a smoking history. The investigators will use the same de-intensification chemoradiotherapy regimen already evaluated in LCCC 1120 and 1413 in patients with HPV-associated OPSCC who have a minimal smoking history and in patients with a smoking history but with wild-type p53. Patients with a smoking history who have mutated p53 will not receive de-intensified chemoradiotherapy, but instead will receive standard doses. The hypothesis is that by using genomics in the patients with a significant smoking history, the investigators will better select those who can be safely de-intensified. Circulating free HPV DNA (cf-HPV-DNA) will also be prospectively assessed from blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age (no upper age limit)
2. T0-3, N0 to N2c, M0 squamous cell carcinoma of the oropharynx
3. Biopsy proven squamous cell carcinoma that is HPV and/or p16 positive
4. Radiologic confirmation of the absence of hematogenous metastasis within 12 weeks prior to treatment
5. ECOG Performance Status 0-1
6. CBC/differential obtained within 8 weeks prior to treatment, with adequate bone marrow function defined as follows: Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl
7. Adequate renal and hepatic function within 4 weeks prior to treatment, defined as follows: Serum creatinine < 2.0 mg/dl; Total bilirubin < 2 x the institutional ULN; AST or ALT < 3 x the institutional ULN
8. Negative pregnancy test within 2 weeks prior to treatment for women of childbearing potential
9. Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment and for 6 weeks following treatment.
10. Patients must be deemed able to comply with the treatment plan and follow-up schedule.
11. Patients must provide study specific informed consent prior to study entry

Exclusion Criteria:

1. Prior history of radiation therapy to the head and neck
2. Prior history of head and neck cancer.
3. Unresectable disease (e.g. immobile node on physical exam, nodal disease that radiographically involves the carotid arteries, nerves)
4. Currently taking Disease Modifying Rheumatoid Drugs (DMRDs)
5. Severe, active co-morbidity, defined as follows: Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; Transmural myocardial infarction within the last 6 months; Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects (Note, however, coagulation parameters are not required for entry into this protocol); Pre-existing ≥ grade 2 neuropathy; Prior organ transplant; Systemic lupus; Psoriatic arthritis
6. Known HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendell Gray Yarbrough, MD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina
  - Rex Healthcare, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chera BS, Kumar S, Shen C, Amdur R, Dagan R, Green R, Goldman E, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Blumberg J, Patel S, Thorp B, Weissler M, Yarbrough W, Sheets N, Mendenhall W, Tan XM, Gupta GP. Plasma Circulating Tumor HPV DNA for the Surveillance of Cancer Recurrence in HPV-Associated Oropharyngeal Cancer. J Clin Oncol. 2020 Apr 1;38(10):1050-1058. doi: 10.1200/JCO.19.02444. Epub 2020 Feb 4. PMID 32017652
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 08/25/2016 through 12/11/2020 at 4 cancer centers in the United States.
Pre-assignment Details: A total of 195 subjects consented and started the study. Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included and 126 subjects with arm/group and follow-up were presented.
Groups:
- Group A: Subjects with oropharyngeal squamous cell carcinoma have more than 10 years of smoking history, without p53 mutation and receiving 60Gy radiotherapy with or without chemotherapy.
- Group B: Subjects with oropharyngeal squamous cell carcinoma have equal to or less than 10 years of smoking history, without p53 mutation and receiving 60Gy radiotherapy with or without chemotherapy
- Group C: Subjects with oropharyngeal squamous cell carcinoma have more than 10 years of smoking history and with the p53 mutation and/or treating physicians' discretion receiving 70Gy radiotherapy with or without chemotherapy.
- Group DataUnknown: Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. Demographic data and site assignment for all subjects were stored centrally. Therefore, arm/group and follow-up data related to sixty-nine subjects are missing.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group DataUnknown
Started | 18 | 105 | 3 | 69
Assessment and Biopsy Was Done if Required at 2 Years After Treatment | 11 | 51 | 2 | 0
Completed | 15 | 100 | 3 | 0
Not Completed | 3 | 5 | 0 | 69
Not completed — Death | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Research at two study sites terminated early | 0 | 0 | 0 | 69

BASELINE CHARACTERISTICS:
Population: Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group data related to sixty-nine subjects are not included in the data tables.
Groups:
- Group Data Unknown: Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. Demographic data and site assignment for all subjects were stored centrally. Therefore, arm/group and follow-up data related to sixty-nine subjects are missing.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group Data Unknown | Total
Number analyzed (Participants) | 18 | 105 | 3 | 69 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.72 (8.43) | 59.89 (9.8) | 61.66 (4.16) | 64.5 (9.74) | 60.86 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 12 | 3 | 3 | 19
  Male | 17 | 93 | 0 | 66 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 16 | 99 | 3 | 67 | 185
  Unknown or Not Reported | 2 | 3 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 1 | 2 | 7
  White | 17 | 91 | 2 | 67 | 177
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 9 | 0 | 0 | 10
Region of Enrollment [Number; unit: participants]
  United States | 18 | 105 | 3 | 69 | 195

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was assessed as the time from the first day of chemoradiation therapy (CRT) until disease progression. Disease progression was defined as biopsy proven tumor cells. Positron emission tomography / computerized tomography (PET/CT) was performed at week 10-16 (optimally at week 12) after completion of therapy. Biopsies were performed for subjects with imaging or clinical exam results suspicious for tumor. Clinical follow-up occurred and chest imaging was performed during the follow-up.
Time Frame: Two years after completion of the treatment
Population: Subjects completed the study procedures including treatment, PET/CT, and biopsy when required, and followed up 2 years after completion of the treatment. Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 51 | 2
Participants
  Biopsy proven relapse was found | 3 | 6 | 0
  Biopsy proven relapse was not found | 8 | 45 | 2

2. Secondary Outcome: Number of Participants With Plasma Circulating Free DNA -Baseline
Description: The number of subjects who have or do not have plasma circulating free Human papillomavirus Deoxyribonucleic acid (HPV- DNA) was tabulated.
Time Frame: Baseline
Population: Subjects started the treatment and provided specimens for plasma circulating free HPV DNA analysis at baseline. Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 63 | 2
Participants
  HPV (+) | 13 | 59 | 2
  HPV (-) | 1 | 4 | 0

3. Secondary Outcome: Number of Participants With Plasma Circulating Free DNA -3months
Description: as for outcome 2
Time Frame: 3 months after completion of the treatment
Population: Subjects completed the study treatment and provided specimens for plasma circulating free HPV DNA analysis at 3 months after the completion of radiotherapy. Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 59 | 1
Participants
  HPV (+) | 3 | 19 | 0
  HPV (-) | 10 | 40 | 1

4. Secondary Outcome: Number of Participants With Plasma Circulating Free DNA -1 Year
Description: as for outcome 2
Time Frame: 1 year after completion of the treatment
Population: Subjects completed the study treatment and provided specimens for plasma circulating free HPV DNA analysis 1 year after the completion of radiotherapy. Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 7 | 51 | 0
Participants
  HPV (+) | 2 | 10 | 0
  HPV (-) | 5 | 41 | 0

5. Secondary Outcome: Number of Participants With Plasma Circulating Free DNA -2 Year
Description: as for outcome 2
Time Frame: 2 years after completion of the treatment
Population: Subjects completed the study treatment and provided specimens for plasma circulating free HPV DNA analysis 2 years after the completion of radiotherapy. Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6 | 39 | 1
Participants
  HPV (+) | 2 | 16 | 0
  HPV (-) | 4 | 23 | 1

6. Secondary Outcome: Local Control Rate
Description: The local control rate is defined as the total disappearance of the primary tumor without any local recurrence. Local recurrence was defined as biopsy-proven tumor cells in the primary tumor region. Biopsy was performed for a subject with a positive positron emission tomography / computerized tomography scan and /or clinical discretion of the surgeon 16 weeks after completion of the treatment.
Time Frame: 2 years after completion of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 51 | 2
Participants
  local relapse | 0 | 0 | 0
  No local relapse | 11 | 51 | 2

7. Secondary Outcome: Regional Control Rate
Description: Regional control rate is defined as the total disease disappearance of the related lymph node metastases without any lymph node recurrence. Regional recurrence was defined as biopsy proven tumor cells in related lymph nodes. Biopsy was performed for a subject with a positive positron emission tomography / computerized tomography scan and /or clinical discretion of the surgeon 16 weeks after completion of the treatment.
Time Frame: 2 years post-CRT
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 51 | 2
Participants
  Biopsy proven regional relapse was found | 1 | 2 | 0
  Biopsy proven regional relapse was not found | 10 | 49 | 2

8. Secondary Outcome: Local-regional Control Rate
Description: Local-regional control rate is defined as the total disappearance of the primary tumor and related lymph node metastases without any recurrence. Local-regional recurrence was defined as biopsy-proven tumor cells in the primary tumor region and/or related lymph nodes. Biopsy was performed for a subject with a positive positron emission tomography / computerized tomography scan and /or clinical discretion of the surgeon 16 weeks after completion of the treatment.
Time Frame: 2 years after completion of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 51 | 2
Participants
  Biopsy proven local or regional relapse was found | 1 | 2 | 0
  Biopsy proven local or regional relapse was not found | 10 | 49 | 2

9. Secondary Outcome: Distant Metastasis Free Survival
Description: Distant metastasis-free survival is defined as the time from the first day of the study treatment to the date of disease spreads while subjects are alive.
  Distant metastasis-free survival is defined as no disease outside of the primary tumor and related lymph node metastases. Distant metastasis was defined as biopsy-proven tumor cells outside of the primary tumor and related lymph node metastases. Biopsy was performed for a subject with a positive positron emission tomography / computerized tomography scan and /or clinical discretion of the surgeon 16 weeks after completion of the treatment.
Time Frame: Two years after completion of the treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 51 | 2
Participants
  Biopsy proven distant metastasis was found | 2 | 4 | 0
  Biopsy proven distant metastasis was not found | 9 | 47 | 2

10. Secondary Outcome: Overall Survival Rate
Description: The overall survival rate is defined as the time from the first day of the study treatment to the date of death for any cause. Subjects who have not had an event will be censored at the date of the last assessment documenting the subject was alive.
Time Frame: Up to 2 years after completion of treatment
Population: Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 12 | 55 | 2
Participants
  Death | 1 | 4 | 0
  Alive | 11 | 51 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Description: The protocol does not require adverse event assessment. Adverse Event Data was not collected.
  Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included.
Groups:
- Group A: Subjects with oropharyngeal squamous cell carcinoma have more than 10 years of smoking history, without p53 mutation and receiving 60Gy radiotherapy with or without chemotherapy.
  Research at two study sites terminated early (halted prematurely due to non-compliance in the performance of the study). Therefore, follow-up data is missing. Data from these subjects is not included in survival calculations.
- Group B: Subjects with oropharyngeal squamous cell carcinoma have equal to or less than 10 years of smoking history, without p53 mutation and receiving 60Gy radiotherapy with or without chemotherapy.
  Research at two study sites terminated early (halted prematurely due to non-compliance in the performance of the study). Therefore, follow-up data is missing. Data from these subjects is not included in survival calculations.
- Group C: Subjects with oropharyngeal squamous cell carcinoma have more than 10 years of smoking history and with the p53 mutation and/or treating physicians' discretion receiving 70Gy radiotherapy with or without chemotherapy.
  Research at two study sites terminated early (halted prematurely due to non-compliance in the performance of the study). Therefore, follow-up data is missing. Data from these subjects is not included in survival calculations.
Arm/Group | Group A | Group B | Group C | Group DataUnknown
All-Cause Mortality (participants affected / at risk) | 1/18 | 4/105 | 0/3 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Research at two study sites terminated early. Each site collected and stored the research data for its participants in its own systems. The validity of existing, sequestered outcome data from sites 3 and 4 cannot be confirmed and may not be reliable. Therefore, arm/group and follow-up data related to sixty-nine subjects are not included in the data tables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LCCC1612 is a multi-site study. Three of the four site investigators are not employees of the Sponsor. Restrictions to disclosure do not apply due to circumstances of non-compliance. Study data was sequestered, data is not accessible for further analysis or publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT03077243/Prot_SAP_000.pdf